CLINICAL TRIAL: NCT03854695
Title: Study to Evaluate Bacterial Activity That Drives the Progression of Clinical Infection
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawing study from PRS-this is not an actual clinical trial
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 052018-055
Record Dates: First submitted 2018-12-10; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 blood samples - one for serum and one collected in PAXgene tubes
  5 tissue samples from wound bed of discarded debridement tissue - one frozen, one fixed in formalin, one placed in RNAlater, one fixed for confocal microscopy and one prepped for Scanning Electron Microscopy (SEM) analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Cohort 1: clinically uninfected (1A and 1C) ulcers.
- Cohort 2: Cohort 2: clinically infected (redness, edema, induration, heat, exudate, tenderness/pain (1B and 1D)) with no recent antibiotic therapy (within 28 days)
- Cohort 3: Cohort 3: clinically infected (redness, edema, induration, heat, exudate, tenderness/pain (1B and 1D)) on antibiotic therapy

SUMMARY:
The investigators plan to enroll up to 750 subjects over the course of 5 years. Study duration will be 2 visits over 7 days (+/-3). Participants will be consented and undergo baseline procedures. Participants will be grouped into 1 of 3 groups, based on infection and antibiotic status at screening. Debridement will be performed per standard of care and collection of tissue will be taken from this discarded tissue. A blood draw will be performed at each of these two visits as well. This is for research purposes only. All other data will be obtained from the electronic medical record. All standard of care except for the blood draws.

DETAILED DESCRIPTION:
Study Groups:

Participants will be divided 1:1:1 into groups with

* Cohort 1: clinically uninfected (1A and 1C) ulcers.
* Cohort 2: clinically infected (redness, edema, induration, heat, exudate, tenderness/pain (1B and 1D)) with no recent antibiotic therapy (within 28 days)
* Cohort 3: clinically infected (redness, edema, induration, heat, exudate, tenderness/pain (1B and 1D)) on antibiotic therapy

Duration of Subject Participation

* Screening: Within 7 days of baseline visit
* Baseline (can be the same day)
* Week 1 visit: one week after baseline.
* Follow-up period - EMR: 6 months from baseline measurements
* Total duration of subject participation: Up to 6 months

Study Procedures:

Screening

1. Explain purpose and nature of the study and obtain signature on the informed consent document and HIPAA Authorization. 2. Screen the subject against protocol inclusion and exclusion criteria, including all pertinent tests.

Baseline (may be done as same day as screening procedures). This visit may last 1.4-2 hours.

1. Obtain general medical history, demographic information and social history.
2. Complete a physical examination of the foot, body weight, height, and vital signs, including measurement of resting heart rate, respiratory rate, and blood pressure while seated.
3. Select the target ulcer.
4. Obtain complete history pertinent to ulcer disease including duration of the target ulcer, previous and current treatment.
5. Perform debridement if indicated. Debridement is to be performed using a curette, scissors, scalpel, or forceps.
6. Obtain study samples a. 2 blood samples - one for serum and one collected in PAXgene tubes b. 5 tissue samples - one frozen, one fixed in formalin, one placed in RNAlater, one fixed for confocal microscopy and one prepped for SEM analysis.
7. Assess the post-debridement ulcer size using a ruler.
8. Perform standardized photography of the study wound.
9. Perform additional vascular and neuropathy studies.
10. Collect all relevant concomitant medications for the previous 28 days.
11. Clinician will perform standard wound care, including wound measurements and photography, and apply appropriate dressings/treatment.
12. Record wound treatment applied including off-loading and debridement.
13. Urine pregnancy test if needed.

Week 1: this visit will not take longer than a normal standard of care visit.

1. Assess target ulcer
2. Debridement is to be performed using curette, scissors, scalpel, or forceps.
3. Obtain study samples a. 2 blood samples - one for serum and one collected in PAXgene tubes b. 5 tissue samples- one frozen, one fixed in formalin, one placed in RNAlater, one fixed for confocal microscopy and one prepped for Scanning Electron Microscopy (SEM) analysis.
4. Perform standard of care wound care per physician discretion including wound measurements and standardized photography of the study wound.
5. Clinician will perform standard wound care, including wound measurements and photography, and apply appropriate dressings/treatment.
6. Record wound treatment applied including off-loading and debridement.
7. Any changes in concomitant medications since baseline will be recorded.
8. Subject stipend disbursement.

Follow up assessment through medical record

1. Wound healing - includes closure or changes in wound size
2. Wound treatment - includes details/changes in treatment regimen.
3. Labs/Concomitant medications/studies related to wound treatment - includes any studies relative to the medical status, wound status, infection, etc.
4. Dehiscence - will be defined as any site along the site of surgical wound closure that fails to have 100% epithelialization without drainage at the time sutures are removed. Often part of the surgical wound will dehisce after it is closed. Therefore, the investigators will evaluate the time until the wound is completely healed. For surgical wounds this will be the time sutures are removed with complete epithelialization of the study wound, or secondary wound healing after previous surgical closure has dehisced.
5. Wound infection - infection will be defined and stratified base in the Infectious Disease Society of Americas classification and criteria.
6. Amputation - The investigators will document amputation using an ordinal scale (no additional amputation, toe and metatarsal, transmetatarsal amputation, midfoot amputation, below the knee, knee disarticulation, and above the knee amputation).
7. Foot related adverse events including hospitalization.
8. The investigators will assess perfusion using Arterial dopplers (bedside may be done for screening if formal ABIs have not yet been performed/resulted) as part of the screening procedures. If other procedures are collected as part of standard of care, those data may be acquired from the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Ankle Brachial Index (ABI) ≥ 0.5 (bedside ABI is acceptable for screening purposes as the formal imaging ABI may not be resulted prior to surgery)

  * One or more chronic lower extremity wounds that are located in the ankle area or below that has persisted a minimum of 30 days prior to the Screening visit, however, only one wound per subject will be included.
  * Ulcer grade I or II, Stage A-D, according to University of Texas Wound Classification System
  * ≥21 years of age or older
  * Diagnosis of diabetes mellitus

Exclusion Criteria:

* • Subject has major immunodeficiency

  * Subject is human immunodeficiency virus (HIV)+
  * Subject has untreated osteomyelitis
  * Subject has active cellulitis
  * Subject has active charcot
  * Is pregnant or plans to become pregnant
  * Is nursing or actively lactating
  * Developmental disability/significant psychological disorder that in the opinion of the investigator could impair the subject's ability to provide informed consent, participate in the study protocol or record study measures, including untreated schizophrenia, bipolar disorder and psychiatric hospitalization within the last 2 years
  * Active alcohol or substance abuse in the opinion of the investigator that could impair the subject's ability to provide informed consent, participate in the study protocol or record study materials

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investgator's patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Assess serum IgG titers | Five years
  Assess serum IgG titers against our target antigens and host gene expression analysis

SECONDARY OUTCOMES:
Characterize microbiology | Five years
  Characterize microbiology (in particular S. aureus) in diabetic foot ulcers (DFU)

OTHER OUTCOMES:
Characterize immune response | Five years
  Characterize microbiology and immune response in DFU biopsy material by confocal microscopy and scanning electron microscopy (UTSW)
Assess microbiome | Five years
  Assess microbiome and the host and bacterial transcriptome in DFU

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, DPM MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States